CLINICAL TRIAL: NCT03986775
Title: AFCRO-066: A Double-blinded, Randomized, Controlled, Acute, Cross-over Study to Determine the Efficacy of Palatinose™ Versus Sucrose on Flow Mediated Dilation in Healthy Subjects With Mild Hypertension
Brief Title: Efficacy of Palatinose™ Versus Sucrose on Flow Mediated Dilation in Healthy Subjects With Mild Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beneo-Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: AFCRO-066
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Overweight and Obesity
Keywords: Glycemic Index; Overweight; Endothelial function; carbohydrate
MeSH Terms: conditions — Overweight; Obesity | interventions — isomaltulose; Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- citrus drink with isomaltulose (Active Comparator)
  Interventions: Dietary Supplement: isomaltulose
- citrus drink with sucrose (Placebo Comparator)
  Interventions: Dietary Supplement: sucrose

INTERVENTIONS:
Dietary Supplement: isomaltulose — replacement of sucrose with low-glycemic isomaltulose
  Arms: citrus drink with isomaltulose
Dietary Supplement: sucrose — conventional beverage with sucrose
  Arms: citrus drink with sucrose

SUMMARY:
To determine the efficacy of Palatinose versus sucrose on Flow Mediated Dilation (FMD) in healthy subjects with mild hypertension.

ELIGIBILITY:
Inclusion criteria:

* Subject is healthy at the time of pre-examination
* Subject has a BMI of 25 - 35 kg/m²
* Subject is aged 25 - 50 years at the time of pre-examination
* Signed written informed consent
* Inactive (IPAQ score <1)
* Waist to Hip ratio ≥0.90 cm for males, ≥0.85 cm for females
* High-normo/Mild hypertensive (SBP: 130-159 mmHg / DBP: 80-99 mmHg)

Exclusion criteria:

* Use of medication interfering with RAAS, such as ACE-inhibitors,
* Advanced cardio-vascular disease (CVD),
* Severe kidney disorders (CKD),
* Diabetes mellitus, both type 1 and II diabetes,
* Pregnant, lactating or wish to become pregnant,
* Hypersensitivity to any of the components of the test product,
* Restricted diet (vegetarian)
* Thyroid disease
* Heavy Smokers (light smokers allowed)
* Lack of suitability for participation in the trial, for any medical reason, as judged by the PI.
* Excessive alcohol consumption (>21 units/week for males & >14 units/week for females)

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-03-03 (Actual); Study Completion 2017-08-09 (Actual)

PRIMARY OUTCOMES:
Brachial ultrasound FMD scan | Baseline, 60 minutes, 120 minutes, 180 minutes
  Changes in postprandial flow-mediated Dilation (endothelial function)

SECONDARY OUTCOMES:
Postprandial glycemic response | Baseline, 60 minutes, 120 minutes, 180 minutes
  Postprandial glycemic response (Plasma samples)
Postprandial insulin response | Baseline, 60 minutes, 120 minutes, 180 minutes
  Postprandial Insulin response (Plasma samples)

IPD SHARING:
Plan to Share IPD: No